CLINICAL TRIAL: NCT07151339
Title: Pilotprojekt Renale Und kardiovaskuläre Tertiärprävention Nach Präeklampsie
Brief Title: Pilot Project Renal and Cardiovascular Tertiary Prevention in Preeclampsia
Acronym: EagleEye3P
Status: Recruiting | Type: Observational
Sponsor: University Hospital Schleswig-Holstein (Other)
Responsible Party: Principal Investigator, Laura Katharina Sievers, Principal Investigator, University Hospital Schleswig-Holstein
Other Study IDs: D557/24
Record Dates: First submitted 2025-08-20; First posted 2025-09-03 (Actual); Last update posted 2025-09-03 (Actual); Status verified 2025-08

CONDITIONS: Preeclampsia; HELLP Syndrome; Eclampsia; Kidney Disease
Keywords: cardiovascular prevention; preeclampsia; pregnancy
MeSH Terms: conditions — Pre-Eclampsia; HELLP Syndrome; Eclampsia; Kidney Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 12 Months
Biospecimen Retention: Samples With DNA — Blood, urine, stool
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Tertiary prevention program for women with preeclampsia, HELLP syndrome, kidney disease and pregnancy or associated conditions, including founding of a biobank. (Observational study since no interference with regular path of treatment suggested in national and international guidelines)

ELIGIBILITY:
Inclusion Criteria:

* older than 18 yrs
* diagnosed preeclampsia, HELLP syndrome or kidney disease durig pregnancy

Exclusion Criteria:

* unable for informed consent

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — women during pregnancy
Study Population: women with preeclampsia/HELLP syndrome/kidney disease during pregnancy
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2024-11-01 (Actual); Primary Completion 2029-11 (Estimated); Study Completion 2030-11 (Estimated)

PRIMARY OUTCOMES:
Pulse wave velocity | 12 months

CONTACTS AND LOCATIONS:
Locations (1):
- University Hospital Schleswig- Holstein, Kiel, Germany

IPD SHARING:
Plan to Share IPD: No